CLINICAL TRIAL: NCT05777148
Title: Comparison of Efficacy in Removal of Advanced Glycation End Products (AGEs) Between Super High-flux Hemodialysis and Postdilution Online Hemodiafiltration: A Single-center, Prospective, Open-label, Crossover Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3619
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: End Stage Renal Disease
Keywords: hemodiafiltration; super high-flux hemodialysis; advanced glycation end products
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postdilution online hemodiafiltration (Experimental): hemodialysis by using post dilution online HDF technique
  Interventions: Device: postdilution online hemodiafiltration
- super high-flux hemodialysis (Experimental): hemodialysis by using super high-flux dialyzer
  Interventions: Device: super high-flux hemodialysis

INTERVENTIONS:
Device: super high-flux hemodialysis — Super high-flux hemodialysis (SHF-HD) is hemodialysis using Super high-flux dialyzer for 24 week then crossover to post dilution online HDF (wash out period 4 weeks)
  Arms: super high-flux hemodialysis
Device: postdilution online hemodiafiltration — hemodialysis by post dilution online HDF technique for 24 week then crossover to super high-flux HD (wash out period 4 weeks)
  Arms: postdilution online hemodiafiltration

SUMMARY:
The goal of this clinical trial is to compare efficacy in advanced glycation end products removal between Super high-flux Hemodialysis and high-volume post-dilution online hemodiafiltration. The main question it aims to answer are

* Efficacy : endothelial dysfunction biomarker (AGEs) in super high-flux hemodialysis compared to online HDF
* Safety profile : Dialysate albumin loss, Intradialytic complication

Participants will be asked to randomized in 2 groups : Super high-flux HD or post dilution ol-HDF Researchers will compare SHF-HD and ol-HDF to see whether SHF-HD could remove AGEs better than ol-HDF

ELIGIBILITY:
Inclusion Criteria:

* Chronic HD > 3 months
* Adequate small molecule uremic toxins removal
* Kt/v > 1.8 in HD 2 times/week
* Kt/v > 1.2 in HD 3 times/week
* BFR > 300 mL/min
* RKF < 100 ml/day
* Hemodynamically stable for > 2 weeks

Exclusion Criteria:

* contraindicated to anticoagulant
* active malignancy
* advanced liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
skin autofluorescence for AGEs | 24 weeks
  SAF was measured by using a certified Autofluorescence Reader (AGE Reader, DiagnOptics, Groningen, The Netherlands). The AGEs reader uses an excitation light source between 300 and 420 nm to illuminate a skin surface that is about 1 cm2 in size and shielded from outside light. A spectrometer (AVS-USB2000, Avantes Inc., Eerbeek, The Netherlands) is used to measure the emission light from the skin in the 300- to 600-nm region using a 200-mm glass fiber.

SECONDARY OUTCOMES:
serum beta 2 microglobulin | At first week, 8th week, 16th week and 24th week
  Measure mid-week prehemodialysis serum beta2 micro globulin

CONTACTS AND LOCATIONS:
Locations (1):
- ramathibodi hospital, faculty of medicine, Ramathibodi hospital, Phaya Thai, Bangkok, Thailand